CLINICAL TRIAL: NCT04746690
Title: Effects of Slider, Tensioner Neurodynamic Mobilization Techniques and Stretching Exercises in Treatment of Chronic Discogenic Sciatica: A Comparative Study
Brief Title: Effects of Neurodynamic Mobilization and Stretching Exercises for Chronic Discogenic Sciatica
Acronym: NDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Ibrahim, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.8/8/93
Record Dates: First submitted 2021-01-31; First posted 2021-02-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Physical Therapy

STUDY DESIGN:
Intervention Model Description: simple random sampling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slider neurodynamic mobilization technique only (Active Comparator): a neurodynamic mobilization technique of the sciatic nerve with stretch on one nerve end and slackness on the other end.
  Interventions: Other: Slider, tensioner neurodynamic mobilization techniques and stretching exercises of back, hamstrings and gastrocnemius
- Tensioner neurodynamic mobilization technique only (Active Comparator): a neurodynamic mobilization technique of the sciatic nerve with stretch of both nerve ends.
  Interventions: Other: Slider, tensioner neurodynamic mobilization techniques and stretching exercises of back, hamstrings and gastrocnemius
- Stretching exercises of back extensors, hamstrings and gastrocnemius muscles (Active Comparator): Stretching exercises of back extensors, hamstrings and gastrocnemius to relief the pressure on the nerve.
  Interventions: Other: Slider, tensioner neurodynamic mobilization techniques and stretching exercises of back, hamstrings and gastrocnemius

INTERVENTIONS:
Other: Slider, tensioner neurodynamic mobilization techniques and stretching exercises of back, hamstrings and gastrocnemius — neurodynamic mobilization techniques of sciatic nerve and stretching exercises of back extensors, hamstrings and lower limbs for patients with chronic discogenic sciatica.
  Other Names: sliders, tensioners and stretching exercise

SUMMARY:
This study compares between neurodynamic mobilization and stretching exercises in treatment of chronic dicogenic sciatica

DETAILED DESCRIPTION:
This study was conducted at the outpatient clinics, faculty of physical Therapy, Kafrelsheikh University to compare between the effects of slider, tensioner neurodynamic mobilization techniques and stretching exercises on pain, Range of motion (ROM) and functional disability for patients with chronic discogenic sciatica.

Design of the study:

A pre-test post-test three-armed comparative study design was used for comparison between the effects of slider, tensioner neurodynamic mobilization techniques and stretching exercises for patients with chronic discogenic sciatica.

Selection of patients:

Sample size:

Using G-power software program and regarding F test study , alpha level of 0.05, confidence interval 95% and effect size of 0.25 (to detect small effects ), three groups and 6 dependent variables, the total sample size will be 36 patient (twelve in each group).

To reach the specific sample size, forty-three patients were screened regarding the inclusion/exclusion criteria. Thirty-six patient with unilateral chronic discogenic sciatica from both sexes (….male and … female) were recruited from the outpatient clinics, faculty of physical Therapy, Kafrelsheikh University. Their age ranged between 21-50 years.

They were randomly allocated by simple random method; to avoid selection bias, patients were asked to choose a card of three wrapped cards representing the three treatment groups:

Group (A): received Slider technique only. Group (B): received Tensioner technique only. Group (C): received Stretching exercises of back extensors, hamstrings and gastrocnemius muscles only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed by magnetic resonance imaging (MRI) confirming disc lesion.
2. Radicular pain for at least twelve weeks up to one year with no acute episodes for the last four weeks.
3. Positive slump test, with reproduction of neurological symptoms.
4. Ages of 21-50 years of both sexes.
5. Patients with functional disabilities e.g. during lifting or walking

Exclusion Criteria:

1. Patients with sciatica due to other pathologies e.g. lumbar canal stenosis or piriformis syndrome.
2. Patients after any spinal surgery e.g. unilateral hemilaminectomy or microdiscectomy
3. Negative slump test.
4. Progressive neurological symptoms e.g. hyperirritable and unstable symptoms.
5. History of vertebral fracture or trauma.
6. Systemic disorder e.g. diabetes mellitus.
7. Pregnant women.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Identity card
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity measurements using visual analogue scale | Before treatment and after 2 weeks of treatment.
  A scale form 0 to 10 points, a less score means improvement.
Change in hip flexion range of motion measurement using universal goniometer. | Before treatment and after 2 weeks of treatment.
  the therapist measures it for patients, an increasing value means improvement.
Change in knee extension range of motion measurement using universal goniometer. | Before treatment and after 2 weeks of treatment.
  the therapist measures it for patients, an increasing value means improvement.
Change in ankle dorsiflexion range of motion measurement using universal goniometer. | Before treatment and after 2 weeks of treatment.
  the therapist measures it for patients, an increasing value means improvement.
Change in lumbar flexion range of motion measurement using universal goniometer. | Before treatment and after 2 weeks of treatment.
  the therapist measures it for patients, an increasing value means improvement.
Change in functional disability measurement using the oswestry disability index. | Before treatment and after 2 weeks of treatment.
  An index indicating disability level, a less score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem El-nahass, Professor, Principal Investigator — Professor of Orthopaedic Physical Therapy
Locations (1):
- Haytham Ibrahim Morsi, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
No availability of participant data